CLINICAL TRIAL: NCT06866665
Title: ADequate AntiPlatelet and Anticoagulation Therapy in Atrial Fibrillation Patients With Focus on Ischemic Risk Management A Randomized ADAPT AFFIRM Study
Brief Title: Antithrombotic Strategy for AF Patients With High Risk CAD
Acronym: ADAPT AFFIRM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2024-1325
Record Dates: First submitted 2025-02-23; First posted 2025-03-10 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation; Coronary Artery Disease
Keywords: Atrial fibrillation; complex PCI; polyvascular disease; antithrombotic strategy
MeSH Terms: conditions — Atrial Fibrillation; Coronary Artery Disease | interventions — Combined Modality Therapy; apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anticoagulation Monotherapy (Active Comparator): Participants receiving anticoagulation monotherapy
  Interventions: Drug: Anticoagulation Monotherapy
- Combination therapy (Experimental): Particiapnts receiving anticoagulation therapy with additional clopidogrel
  Interventions: Drug: Combination therapy

INTERVENTIONS:
Drug: Anticoagulation Monotherapy — Participants in the anticoagulation monotherapy group will receive apixaban 5 mg twice daily during the study period.
  Other Names: Apixaban monotherapy
  Arms: Anticoagulation Monotherapy
Drug: Combination therapy — Participants in the combination therapy group will receive clopiogrel 75 mg daily and apixaban 5 mg twice daily during the study period.
  Other Names: Apixaban and clopidogrel combination therapy
  Arms: Combination therapy

SUMMARY:
Anticoagulation therapy is recommended for patients with atrial fibrillation (AF) in order to prevent ischemic stroke and systemic embolism. Meanwhile, lifelong antiplatelet therapy is highly recommended to prevent stent thrombosis and further ischemic adverse events after percutaneous coronary intervention (PCI) with drug-eluting stent (DES) implantation. In this context, in patients with AF undergoing DES implantation, anticoagulation and antiplatelet therapies perform their own unique roles. However, the current guidelines recommend to discontinue this antiplatelet agent beyond 1 year due to an excessive bleeding risk derived from DAT.

The Atrial Fibrillation and Ischemic Events with Rivaroxaban in Patients with Stable Coronary Artery Disease (AFIRE) emphasized that bleeding risk derived from rivaroxaban-based DAT may outweigh ischemic risk derived from antiplatelet discontinuation in patients with AF and stable coronary artery disease. Furthermore, the recent Edoxaban versus Edoxaban with Antiplatelet Agent in Patients with Atrial Fibrillation and Chronic Stable Coronary Artery Disease (EPIC-CAD) trial also demonstrated that edoxaban monotherapy led to a lower net adverse event compared to than edoxaban-based DAT.

Although these studies strongly supported the benefit of antiplatelet discontinuation in AF patients with stable coronary artery disease, many physicians still hesitate to discontinue antiplatelet agents even 1 year after DES implantation because of concerns regarding stent thrombosis or subsequent myocardial infarction (MI). This concern is exacerbated in patients with an excessive ischemic risk, such as those who received complex PCI or those with polyvascular disease. To address this disparity between clinical practice and recommendations based on the guidelines, the Adequate Antiplatelet and Anticoagulation Therapy in Atrial Fibrillation Patients with Focus on Ischemic Risk Management (ADAPT AFFIRM) trial is designed to elucidate the efficacy and safety of apixaban monotherapy versus apixaban plus clopidogrel combination therapy as a chronic maintenance strategy in AF patients with stable coronary artery disease and excessive ischemic risk.

DETAILED DESCRIPTION:
Investigators will recruit 1400 patients with atrial fibrillation (AF) and coronary artery disease (CAD) with high ischemic risk. High ischemic risk is defined as acute myocardial infarction, complex percutaneous coronary intervention (PCI), untreated significant coronary stenosis, or polyvascular disease. Paticipants will be randomly assigned to either anticoagulation monotherapy group or combination therapy group. Participants assigned to the anticoagulation monotherapy group wil receive apixaban 5 mg twice daily (or reduced dose as judged by investigators) and those assigned to the combination therapy group will receive additional clopidogrel 75 mg daily on top of apixaban. Net adverse clinical events comprising all-cause death, myocardial infarction, stroke, systemic embolism, or ISTH major or clinically relevant non-major bleeding events will be evaluated at 12 months after randomization. Included participant will be followed up until the last participant will be followed up for at lease 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 19 years old
2. Presence of AF with CHA2DS2-VASc score ≥ 2
3. Patients with stable CAD - a history of percutaneous coronary intervention (PCI) or coronary artery bypass graft surgery (CABG) before 6 months (chronic coronary syndrome) or 12 months (acute coronary syndrome); anatomically confirmed CAD on coronary angiography or computed tomography scan
4. Presence of an excessive ischemic risk i. A history of myocardial infarction (MI) ii. Complex PCI iii. Untreated lesion with >50% stenosis at major epicardial vessel after coronary revascularization iv. Untreated multivessel CAD (>50% stenosis of >1 major epicardial vessel or left main stem) v. Peripheral artery disease vi. Cerebrovascular disease

Exclusion Criteria:

1. >85 years old.
2. Patients who received PCI or CABG within 6 months.
3. Patients with a history of acute coronary syndrome within 12 months.
4. Patients who require anticoagulation with warfarin due to a mechanical prosthetic valve, or ≥ moderate mitral stenosis.
5. Patients with a comorbidity requiring anticoagulation other than AF.
6. Patients who is not able to receive apixaban or clopidogrel due to previous adverse reaction.
7. Patients who have coagulopathy or have a history of recurrent bleeding.
8. Intracranial or gastrointestinal bleeding within 3 months.
9. Gastrointestinal tumor requiring treatment.
10. Patients who are pregnant or those who report potential pregnancy.
11. Life expectancy < 1 year due to malignancy.
12. Refuse or enable to understand the written informed consent.
13. Patiens who are not able to discontinue a drug related to CYP3A4 inhibition.

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Net adverse clinical event (NACE) | 12 months after the last enrollment
  NACE is defined as a composite of all-cause death, MI, stroke, systemic embolism, and major or clinically relevant non-major (CRNM) bleeding as defined by International Society on Thrombosis and Hemostasis (ISTH) criteria.

SECONDARY OUTCOMES:
Composite bleeding event | 12 months after the last enrollment
  Composite bleeding event: a composite of ISTH major or CRNM bleeding
Major adverse cardiac event | 12 months after the last enrollment
  Major adverse cardiac event (MACE): a composite of cardiovascular death, MI, or any coronary revascularization
Key ischemic event | 12 months after the last enrollment
  Key ischemic event: a composite of cardiovascular death, MI, ischemic stroke, or systemic embolism
Each components of NACE | 12 months after the last enrollment
  all-cause death
Cardiovascular death | 12 months after the last enrollment
Non-cardiovascular death | 12 months after the last enrollment
Ischemic stroke | 12 months after the last enrollment
Hemorrhagic stroke | 12 months after the last enrollment
Any coronary revascularization | 12 months after the last enrollment
  PCI (Percutaneous Coronary Intervention), CABG(Coronary Artery Bypass Graft)
Acute limb ischemia | 12 months after the last enrollment
Any limb revascularization or amputation | 12 months after the last enrollment
  1. Endovascular revascularization
  2. Surgical revascularization
  3. Amputation
Any intracranial revascularization | 12 months after the last enrollment
  1. Endovascular revascularization
  2. Surgical revascularization
A composite of cardiovascular death, MI, acute limb ischemic, or any limb revascularization or amputation | 12 months after the last enrollment
A composite of cardiovascular death, MI, acute limb ischemia, or ischemic stroke | 12 months after the last enrollment
Each components of NACE | 12 months after the last enrollment
  stroke
Each components of NACE | 12 months after the last enrollment
  systemic embolism
Each components of NACE | 12 months after the last enrollment
  ISTH major bleeding
Each components of NACE | 12 months after the last enrollment
  ISTH CRNM bleeding
Each components of NACE | 12 months after the last enrollment
  MI

IPD SHARING:
Plan to Share IPD: Undecided